CLINICAL TRIAL: NCT05747144
Title: Multimodal Imaging in Vitreo-retinal Surgery and Macular Dystrophies: Biomarkers of Morpho-Functional Recovery by Artificial Intelligence
Brief Title: Multimodal Imaging in Vitreo-retinal Surgery and Macular Dystrophies
Acronym: MICAI
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RIZZO STANISLAO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3680
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Macular Holes; Epiretinal Membrane; Retinal Detachment; Macular Dystrophies
Keywords: vitreoretinal surgery; machine learning; decisional support systems
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane; Retinal Detachment; Macular Degeneration | interventions — Color

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Macular hole: Patients affected by macular hole.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Retinography (Color) + Autofluorescence (AF); Diagnostic Test: OCT B-scan and OCT angiography (OCTA); Diagnostic Test: Microperimetry; Diagnostic Test: Electrophysiological exams
- Epiretinal membranes: Patients affected by epiretinal membrane.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Retinography (Color) + Autofluorescence (AF); Diagnostic Test: OCT B-scan and OCT angiography (OCTA); Diagnostic Test: Microperimetry; Diagnostic Test: Electrophysiological exams
- Retinal detachment: Patients affected by retinal detachment.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Retinography (Color) + Autofluorescence (AF); Diagnostic Test: OCT B-scan and OCT angiography (OCTA); Diagnostic Test: Microperimetry; Diagnostic Test: Electrophysiological exams
- Macular dystrophies: Patients affected by macular dystrophies.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Retinography (Color) + Autofluorescence (AF); Diagnostic Test: OCT B-scan and OCT angiography (OCTA); Diagnostic Test: Microperimetry; Diagnostic Test: Electrophysiological exams

INTERVENTIONS:
Diagnostic Test: Biometry — Biometric measurements performed with IOL Master, if executable Contact or immersion echobiometry if IOL Master cannot be performed
Diagnostic Test: Retinography (Color) + Autofluorescence (AF) — Colour + AF: EIDON, if available (60° not modulable) Colour: COBRA (60° non-modifiable) AF: Spectralis-Heidelberg (choose 55°) Other if available (choose posterior pole examination between 50-60°)
Diagnostic Test: OCT B-scan and OCT angiography (OCTA) — OCT B-scan:
  2 scans (6 mm)
  1 cross line
  OCTA:
  3x3 mm + 6x6 mm centred on the fovea 4.5 mm centred on the optic nerve
Diagnostic Test: Microperimetry — 1) fixation pattern 2) retinal sensitivity map
Diagnostic Test: Electrophysiological exams — Layer-by-layer assessment of the retina using focal ERG and pattern ERG according to standardised and published methods , For patients with visus < 3/10 and unstable fixation a protocol based on component analysis of the photopic ERG from diffuse flash will be used.

SUMMARY:
The aim of the study is to identify morphological and functional biomarkers of post-operative recovery after vitreoretinal surgery, using decisional support systems (DSS), based on multimodal big-data analysis by means of machine learning techniques in daily clinical practice

DETAILED DESCRIPTION:
The aim of the study is to identify morphological and functional biomarkers of post-operative recovery after vitreoretinal surgery. Identifying the biomarkers and assessing the predictivity of recovery will make it possible to highlight the categories of patients who can benefit most from surgical treatment, and to target the patient more precisely for personalised medicine and surgery. The introduction of new decisional support systems (DSS), based on multimodal big-data analysis through machine learning techniques in daily clinical practice, is providing new useful information in patient assessment for personalised surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients to undergo vitreo-retinal surgery for:

  1. Macular hole
  2. Epiretinal membranes
  3. Retinal detachment
  4. Macular dystrophies (retinal pre-prosthesis)

Exclusion Criteria:

* Patients under 18 years of age will be excluded; patients in whom morphological examinations cannot be performed due to poor cooperation or opacity of the dioptric media (e.g. corneal pathology). Quality of morphological images inadequate for post acquisition processing (<6/10).

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients to undergo vitreo-retinal surgery for macular disease (i.e.Macular hole, epiretinal membranes, Retinal detachment, Macular dystrophies (retinal pre-prosthesis).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-16 (Estimated)

PRIMARY OUTCOMES:
Predictivity of morphological-functional radiomic data | 3 years
  Rate of predictivity of morphological-functional radiomic data to establish the grade of recovery in the post-operative period by means of an artificial intelligence (AI) machine learning model.

SECONDARY OUTCOMES:
Identify predictive differences according to diagnosis | 3 years
  Subdivision into subgroups in order to identify predictive differences according to diagnosis
Correlating with the age of patients | 3 years
  Identify predictive differences according to diagnosis and correlate them with the age of patients
Correlate with age of onset of disease | 3 years
  Identify predictive differences according to diagnosis and correlate them with the age of onset of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Stanislao Rizzo, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garrity ST, Sarraf D, Freund KB, Sadda SR. Multimodal Imaging of Nonneovascular Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2018 Mar 20;59(4):AMD48-AMD64. doi: 10.1167/iovs.18-24158. PMID 30025107
- [Background] Acon D, Wu L. Multimodal Imaging in Diabetic Macular Edema. Asia Pac J Ophthalmol (Phila). 2018 Jan-Feb;7(1):22-27. doi: 10.22608/APO.2017504. Epub 2017 Jan 29. PMID 29376234
- [Background] Duker JS, Kaiser PK, Binder S, de Smet MD, Gaudric A, Reichel E, Sadda SR, Sebag J, Spaide RF, Stalmans P. The International Vitreomacular Traction Study Group classification of vitreomacular adhesion, traction, and macular hole. Ophthalmology. 2013 Dec;120(12):2611-2619. doi: 10.1016/j.ophtha.2013.07.042. Epub 2013 Sep 17. PMID 24053995
- [Background] Spaide RF, Fujimoto JG, Waheed NK, Sadda SR, Staurenghi G. Optical coherence tomography angiography. Prog Retin Eye Res. 2018 May;64:1-55. doi: 10.1016/j.preteyeres.2017.11.003. Epub 2017 Dec 8. PMID 29229445
- [Background] Sun P, Tandias RM, Yu G, Arroyo JG. SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY FINDINGS AND VISUAL OUTCOME AFTER TREATMENT FOR VITREOMACULAR TRACTION. Retina. 2019 Jun;39(6):1054-1060. doi: 10.1097/IAE.0000000000002116. PMID 29595569
- [Background] Lee CS, Tyring AJ, Deruyter NP, Wu Y, Rokem A, Lee AY. Deep-learning based, automated segmentation of macular edema in optical coherence tomography. Biomed Opt Express. 2017 Jun 23;8(7):3440-3448. doi: 10.1364/BOE.8.003440. eCollection 2017 Jul 1. PMID 28717579
- [Background] Zur D, Iglicki M, Busch C, Invernizzi A, Mariussi M, Loewenstein A; International Retina Group. OCT Biomarkers as Functional Outcome Predictors in Diabetic Macular Edema Treated with Dexamethasone Implant. Ophthalmology. 2018 Feb;125(2):267-275. doi: 10.1016/j.ophtha.2017.08.031. Epub 2017 Sep 19. PMID 28935399
- [Background] Beam AL, Kohane IS. Big Data and Machine Learning in Health Care. JAMA. 2018 Apr 3;319(13):1317-1318. doi: 10.1001/jama.2017.18391. No abstract available. PMID 29532063
- [Background] Ngiam KY, Khor IW. Big data and machine learning algorithms for health-care delivery. Lancet Oncol. 2019 May;20(5):e262-e273. doi: 10.1016/S1470-2045(19)30149-4. PMID 31044724
- [Background] Abramoff MD, Lou Y, Erginay A, Clarida W, Amelon R, Folk JC, Niemeijer M. Improved Automated Detection of Diabetic Retinopathy on a Publicly Available Dataset Through Integration of Deep Learning. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5200-5206. doi: 10.1167/iovs.16-19964. PMID 27701631
- [Background] Gulshan V, Peng L, Coram M, Stumpe MC, Wu D, Narayanaswamy A, Venugopalan S, Widner K, Madams T, Cuadros J, Kim R, Raman R, Nelson PC, Mega JL, Webster DR. Development and Validation of a Deep Learning Algorithm for Detection of Diabetic Retinopathy in Retinal Fundus Photographs. JAMA. 2016 Dec 13;316(22):2402-2410. doi: 10.1001/jama.2016.17216. PMID 27898976
- [Background] Lakhani P, Sundaram B. Deep Learning at Chest Radiography: Automated Classification of Pulmonary Tuberculosis by Using Convolutional Neural Networks. Radiology. 2017 Aug;284(2):574-582. doi: 10.1148/radiol.2017162326. Epub 2017 Apr 24. PMID 28436741
- [Background] Esteva A, Kuprel B, Novoa RA, Ko J, Swetter SM, Blau HM, Thrun S. Dermatologist-level classification of skin cancer with deep neural networks. Nature. 2017 Feb 2;542(7639):115-118. doi: 10.1038/nature21056. Epub 2017 Jan 25. PMID 28117445
- [Background] Ting DSW, Cheung CY, Lim G, Tan GSW, Quang ND, Gan A, Hamzah H, Garcia-Franco R, San Yeo IY, Lee SY, Wong EYM, Sabanayagam C, Baskaran M, Ibrahim F, Tan NC, Finkelstein EA, Lamoureux EL, Wong IY, Bressler NM, Sivaprasad S, Varma R, Jonas JB, He MG, Cheng CY, Cheung GCM, Aung T, Hsu W, Lee ML, Wong TY. Development and Validation of a Deep Learning System for Diabetic Retinopathy and Related Eye Diseases Using Retinal Images From Multiethnic Populations With Diabetes. JAMA. 2017 Dec 12;318(22):2211-2223. doi: 10.1001/jama.2017.18152. PMID 29234807
- [Background] Li Z, He Y, Keel S, Meng W, Chang RT, He M. Efficacy of a Deep Learning System for Detecting Glaucomatous Optic Neuropathy Based on Color Fundus Photographs. Ophthalmology. 2018 Aug;125(8):1199-1206. doi: 10.1016/j.ophtha.2018.01.023. Epub 2018 Mar 2. PMID 29506863
- [Background] Burlina P, Joshi N, Pacheco KD, Freund DE, Kong J, Bressler NM. Utility of Deep Learning Methods for Referability Classification of Age-Related Macular Degeneration. JAMA Ophthalmol. 2018 Nov 1;136(11):1305-1307. doi: 10.1001/jamaophthalmol.2018.3799. PMID 30193354
- [Background] Grassmann F, Mengelkamp J, Brandl C, Harsch S, Zimmermann ME, Linkohr B, Peters A, Heid IM, Palm C, Weber BHF. A Deep Learning Algorithm for Prediction of Age-Related Eye Disease Study Severity Scale for Age-Related Macular Degeneration from Color Fundus Photography. Ophthalmology. 2018 Sep;125(9):1410-1420. doi: 10.1016/j.ophtha.2018.02.037. Epub 2018 Apr 10. PMID 29653860
- [Background] Brown JM, Campbell JP, Beers A, Chang K, Ostmo S, Chan RVP, Dy J, Erdogmus D, Ioannidis S, Kalpathy-Cramer J, Chiang MF; Imaging and Informatics in Retinopathy of Prematurity (i-ROP) Research Consortium. Automated Diagnosis of Plus Disease in Retinopathy of Prematurity Using Deep Convolutional Neural Networks. JAMA Ophthalmol. 2018 Jul 1;136(7):803-810. doi: 10.1001/jamaophthalmol.2018.1934. PMID 29801159
- [Background] Kermany DS, Goldbaum M, Cai W, Valentim CCS, Liang H, Baxter SL, McKeown A, Yang G, Wu X, Yan F, Dong J, Prasadha MK, Pei J, Ting MYL, Zhu J, Li C, Hewett S, Dong J, Ziyar I, Shi A, Zhang R, Zheng L, Hou R, Shi W, Fu X, Duan Y, Huu VAN, Wen C, Zhang ED, Zhang CL, Li O, Wang X, Singer MA, Sun X, Xu J, Tafreshi A, Lewis MA, Xia H, Zhang K. Identifying Medical Diagnoses and Treatable Diseases by Image-Based Deep Learning. Cell. 2018 Feb 22;172(5):1122-1131.e9. doi: 10.1016/j.cell.2018.02.010. PMID 29474911
- [Background] De Fauw J, Ledsam JR, Romera-Paredes B, Nikolov S, Tomasev N, Blackwell S, Askham H, Glorot X, O'Donoghue B, Visentin D, van den Driessche G, Lakshminarayanan B, Meyer C, Mackinder F, Bouton S, Ayoub K, Chopra R, King D, Karthikesalingam A, Hughes CO, Raine R, Hughes J, Sim DA, Egan C, Tufail A, Montgomery H, Hassabis D, Rees G, Back T, Khaw PT, Suleyman M, Cornebise J, Keane PA, Ronneberger O. Clinically applicable deep learning for diagnosis and referral in retinal disease. Nat Med. 2018 Sep;24(9):1342-1350. doi: 10.1038/s41591-018-0107-6. Epub 2018 Aug 13. PMID 30104768
- [Background] Schmidt-Erfurth U, Sadeghipour A, Gerendas BS, Waldstein SM, Bogunovic H. Artificial intelligence in retina. Prog Retin Eye Res. 2018 Nov;67:1-29. doi: 10.1016/j.preteyeres.2018.07.004. Epub 2018 Aug 1. PMID 30076935
- [Background] Schmidt-Erfurth U, Waldstein SM, Klimscha S, Sadeghipour A, Hu X, Gerendas BS, Osborne A, Bogunovic H. Prediction of Individual Disease Conversion in Early AMD Using Artificial Intelligence. Invest Ophthalmol Vis Sci. 2018 Jul 2;59(8):3199-3208. doi: 10.1167/iovs.18-24106. PMID 29971444
- [Background] Sarao V, Veritti D, Borrelli E, Sadda SVR, Poletti E, Lanzetta P. A comparison between a white LED confocal imaging system and a conventional flash fundus camera using chromaticity analysis. BMC Ophthalmol. 2019 Nov 19;19(1):231. doi: 10.1186/s12886-019-1241-8. PMID 31744471
- [Background] Fernandez-Avellaneda P, Breazzano MP, Fragiotta S, Xu X, Zhang Q, Wang RK, Freund KB. BACILLARY LAYER DETACHMENT OVERLYING REDUCED CHORIOCAPILLARIS FLOW IN ACUTE IDIOPATHIC MACULOPATHY. Retin Cases Brief Rep. 2022 Jan 1;16(1):59-66. doi: 10.1097/ICB.0000000000000943. PMID 31764886
- [Background] Huang NT, Georgiadis C, Gomez J, Tang PH, Drayna P, Koozekanani DD, van Kuijk FJGM, Montezuma SR. Comparing fundus autofluorescence and infrared imaging findings of peripheral retinoschisis, schisis detachment, and retinal detachment. Am J Ophthalmol Case Rep. 2020 Mar 26;18:100666. doi: 10.1016/j.ajoc.2020.100666. eCollection 2020 Jun. PMID 32258825
- [Background] Stanga PE, Williams JI, Shaarawy SA, Agarwal A, Venkataraman A, Kumar DA, You TT, Hope RS. FIRST-IN-HUMAN CLINICAL STUDY TO INVESTIGATE THE EFFECTIVENESS AND SAFETY OF PARS PLANA VITRECTOMY SURGERY USING A NEW HYPERSONIC TECHNOLOGY. Retina. 2020 Jan;40(1):16-23. doi: 10.1097/IAE.0000000000002365. PMID 30358763
- [Background] Hubschman JP, Govetto A, Spaide RF, Schumann R, Steel D, Figueroa MS, Sebag J, Gaudric A, Staurenghi G, Haritoglou C, Kadonosono K, Thompson JT, Chang S, Bottoni F, Tadayoni R. Optical coherence tomography-based consensus definition for lamellar macular hole. Br J Ophthalmol. 2020 Dec;104(12):1741-1747. doi: 10.1136/bjophthalmol-2019-315432. Epub 2020 Feb 27. PMID 32107208
- [Background] Bae K, Lee SM, Kang SW, Kim ES, Yu SY, Kim KT. Atypical epiretinal tissue in full-thickness macular holes: pathogenic and prognostic significance. Br J Ophthalmol. 2019 Feb;103(2):251-256. doi: 10.1136/bjophthalmol-2017-311810. Epub 2018 Apr 26. PMID 29699982
- [Background] Rizzo S, Tartaro R, Barca F, Caporossi T, Bacherini D, Giansanti F. INTERNAL LIMITING MEMBRANE PEELING VERSUS INVERTED FLAP TECHNIQUE FOR TREATMENT OF FULL-THICKNESS MACULAR HOLES: A COMPARATIVE STUDY IN A LARGE SERIES OF PATIENTS. Retina. 2018 Sep;38 Suppl 1:S73-S78. doi: 10.1097/IAE.0000000000001985. PMID 29232338
- [Background] Christensen UC. Value of internal limiting membrane peeling in surgery for idiopathic macular hole and the correlation between function and retinal morphology. Acta Ophthalmol. 2009 Dec;87 Thesis 2:1-23. doi: 10.1111/j.1755-3768.2009.01777.x. PMID 19912135
- [Background] Fukuyama H, Ishikawa H, Komuku Y, Araki T, Kimura N, Gomi F. Comparative analysis of metamorphopsia and aniseikonia after vitrectomy for epiretinal membrane, macular hole, or rhegmatogenous retinal detachment. PLoS One. 2020 May 8;15(5):e0232758. doi: 10.1371/journal.pone.0232758. eCollection 2020. PMID 32384099
- [Background] Rizzo S, Savastano A, Bacherini D, Savastano MC. Vascular Features of Full-Thickness Macular Hole by OCT Angiography. Ophthalmic Surg Lasers Imaging Retina. 2017 Jan 1;48(1):62-68. doi: 10.3928/23258160-20161219-09. PMID 28060396
- [Background] Bacherini D, Savastano MC, Dragotto F, Finocchio L, Lenzetti C, Bitossi A, Tartaro R, Giansanti F, Barca F, Savastano A, Caporossi T, Vannozzi L, Sodi A, Luca M, Faraldi F, Virgili G, Rizzo S. Morpho-Functional Evaluation of Full-Thickness Macular Holes by the Integration of Optical Coherence Tomography Angiography and Microperimetry. J Clin Med. 2020 Jan 15;9(1):229. doi: 10.3390/jcm9010229. PMID 31952306
- [Background] Qi Y, Wang Z, Li SM, You Q, Liang X, Yu Y, Liu W. Effect of internal limiting membrane peeling on normal retinal function evaluated by microperimetry-3. BMC Ophthalmol. 2020 Apr 9;20(1):140. doi: 10.1186/s12886-020-01383-3. PMID 32272972
- [Background] Smith AJ, Telander DG, Zawadzki RJ, Choi SS, Morse LS, Werner JS, Park SS. High-resolution Fourier-domain optical coherence tomography and microperimetric findings after macula-off retinal detachment repair. Ophthalmology. 2008 Nov;115(11):1923-9. doi: 10.1016/j.ophtha.2008.05.025. Epub 2008 Jul 31. PMID 18672289
- [Background] Reumueller A, Wassermann L, Salas M, Karantonis MG, Sacu S, Georgopoulos M, Drexler W, Pircher M, Pollreisz A, Schmidt-Erfurth U. Morphologic and Functional Assessment of Photoreceptors After Macula-Off Retinal Detachment With Adaptive-Optics OCT and Microperimetry. Am J Ophthalmol. 2020 Jun;214:72-85. doi: 10.1016/j.ajo.2019.12.015. Epub 2019 Dec 25. PMID 31883465
- [Background] Falsini B, Serrao S, Fadda A, Iarossi G, Porrello G, Cocco F, Merendino E. Focal electroretinograms and fundus appearance in nonexudative age-related macular degeneration. Quantitative relationship between retinal morphology and function. Graefes Arch Clin Exp Ophthalmol. 1999 Mar;237(3):193-200. doi: 10.1007/s004170050218. PMID 10090581
- [Background] Falsini B, Bardocci A, Porciatti V, Bolzani R, Piccardi M. Macular dysfunction in multiple sclerosis revealed by steady-state flicker and pattern ERGs. Electroencephalogr Clin Neurophysiol. 1992 Jan;82(1):53-9. doi: 10.1016/0013-4694(92)90182-h. PMID 1370144
- [Background] Abed E, Placidi G, Campagna F, Federici M, Minnella A, Guerri G, Bertelli M, Piccardi M, Galli-Resta L, Falsini B. Early impairment of the full-field photopic negative response in patients with Stargardt disease and pathogenic variants of the ABCA4 gene. Clin Exp Ophthalmol. 2018 Jul;46(5):519-530. doi: 10.1111/ceo.13115. Epub 2017 Dec 28. PMID 29178665
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Derived] Savastano MC, Carla MM, Giannuzzi F, Fossataro C, Cestrone V, Boselli F, Biagini I, Beccia F, Raffaele Q, Gravina G, Rizzo C, Savastano A, Rizzo S. OCT analysis of preoperative foveal microstructure in recent-onset macula-off rhegmatogenous retinal detachment: visual acuity prognostic factors. Br J Ophthalmol. 2024 Nov 22;108(12):1743-1748. doi: 10.1136/bjo-2024-325278. PMID 38719346